CLINICAL TRIAL: NCT00283205
Title: Yoga for Treatment of Hot Flashes and Menopausal Symptoms
Brief Title: Yoga for Treatment of Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H5287-26599
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Menopause-related Hot Flashes
Keywords: Menopausal Symptoms; Hot Flashes; Yoga
MeSH Terms: conditions — Hot Flashes | interventions — Yoga

INTERVENTIONS:
Behavioral: Yoga

SUMMARY:
The Yoga for Treatment of Hot Flashes and Menopausal Symptoms is an uncontrolled pilot clinical trial to determine the feasibility of recruitment and of evaluating yoga for the relief of menopausal hot flashes in 12 peri- or postmenopausal women. Participants will attend an Introductory Yoga Workshop, 8 yoga training sessions in 8 weeks, be assessed clinically before, during, and after training and contacted by telephone 3 months later.

DETAILED DESCRIPTION:
This is an uncontrolled pilot trial of yoga among 12 healthy peri- or postmenopausal women experiencing at least 4 hot flashes per day or 30 hot flashes per week. Participants will complete a Screening and Baseline Visit, and then be taught yoga during weekly sessions that will be held in the evening at the Laurel Heights Conference Center. The yoga postures and breathing techniques will be taught by a qualified and certified yoga instructor using the standardized protocol determined by a Yoga Expert Panel. Each group yoga session will take approximately 90 minutes. Participants will also be required to practice yoga at home at least 3 times per week, and be given yoga materials (mat, blocks, straps), and an instruction manual for their use at home. They will be asked to keep a calendar log of the dates/times that they practiced yoga at home. Outcomes will be assessed midway through the yoga training and at a Final Visit.

The main efficacy outcomes are change in number of hot flashes per week and change in severity of hot flashes from baseline to post-training reported on a 7-day diary. We will also measure changes in sleep and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Self-report ≥4 moderate to severe hot flashes per day or ≥ 30 moderate to severe hot flashes per week.
2. Successful completion of a Hot Flash Diary.
3. Able and willing to attend yoga training sessions, maintain yoga logs, and practice yoga at home.

Exclusion Criteria:

1. Inability to sign an informed consent or fill out questionnaires.
2. Use of other treatments for hot flashes (estrogens, progestins, clonidine, selective serotonin reuptake inhibitors,relaxation techniques or acupuncture) within 4 weeks of enrollment in the trial and do not agree to refrain from using these therapies for the duration of the trial.
3. Use of raloxifene or tamoxifen within three months of enrollment.
4. Any condition that, in the investigator's opinion, would preclude the participant from being able to understand and follow the yoga training or from completing the trial, including severe illness, plans to move, substance abuse, significant psychiatric problems, or dementia.

   -

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-09; Study Completion 2005-12

PRIMARY OUTCOMES:
Reduction of number and severity of hot flashes will be summarized by the sample averages.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Grady, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Women's Health Clinical Research Center, San Francisco, California, United States